CLINICAL TRIAL: NCT07226011
Title: Accelerated High-Dose tDCS for Depression: An Open-Label Outpatient Pilot Study
Brief Title: Accelerated High-Dose tDCS for Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark George, Distinguished University Professor of Psychiatry, Radiology and Neuroscience, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00146983; R25DA020537 (NIH)
Record Dates: First submitted 2025-11-04; First posted 2025-11-10 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Major Depression; Major Depression Disorders
Keywords: Depression; Nervous System; tDCS; Interventional; Brain Stimulation; Transcranial Direct Stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Neurologic Manifestations | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The model will include a safety run-in with the first 3 patients, to ensure there are no serious side effects to the dose escalation from 2 mA to 6 mA before enrolling the remaining participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Experimental: High-Dose tDCS Intervention (Experimental): Participants in this single-arm, open-label pilot study will receive high-dose transcranial direct current stimulation (tDCS) for major depressive disorder. Each participant undergoes twice-daily 20-minute sessions at 6 mA for five consecutive weekdays (total of 10 sessions).
  The first three participants complete an in-lab dose-escalation safety run-in (2 mA → 4 mA → 6 mA on Day 1) with a Day 2 skin integrity check before continuing at 6 mA twice daily for the remaining days.
  All participants complete baseline, post-intervention, and 4-week follow-up assessments of depressive symptoms, cognition, and tolerability.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Participants receive transcranial direct current stimulation (tDCS) using a high-dose (6 mA) protocol delivered twice daily for five consecutive weekdays (10 sessions total). The first three participants complete a Day 1 in-lab dose-escalation (2 mA → 4 mA → 6 mA) with a Day 2 skin integrity check before continuing at 6 mA. All sessions last 20 minutes and are followed by adverse-event monitoring.

SUMMARY:
In this study, investigators are testing whether a higher dose of a non-invasive brain stimulation technique, called transcranial direct current stimulation (tDCS), can be safely used in people with depression. Participants will come to the Brain Stimulation Lab and receive mild electrical stimulation through electrodes placed on their scalp.

The study begins with a safety run-in, where the first few participants will receive stimulation at gradually increasing levels (2, 4, and 6 milliamps) while being closely monitored. If no serious side effects are found, later participants will receive repeated 6 milliamp sessions for 5 days total. Investigators will check skin comfort, mood, and overall tolerability after each session.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) remains one of the leading causes of disability worldwide, with many patients experiencing inadequate response to currently available treatments. Transcranial direct current stimulation (tDCS) has shown promise as a non-invasive, well-tolerated neuromodulation technique for depression, but nearly all prior studies have used lower current intensities (≤2 mA). Preliminary modeling and experimental work suggest that higher current dosing may be necessary to achieve sufficient engagement of cortical targets and produce stronger clinical effects.

The present study is designed to address this gap by systematically evaluating the safety, tolerability, and feasibility of high-dose tDCS delivered at 6 mA in adults with MDD. Establishing safety at this higher intensity is a critical step before pursuing larger efficacy trials. By carefully monitoring adverse events and skin integrity during an initial run-in phase, this study provides an evidence base for whether 6 mA tDCS can be safely implemented in a clinical population.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70.
* Current MDD diagnosis (MINI v7).
* Baseline PHQ-9 > 9.
* Capacity to consent
* Fluent English.

Exclusion Criteria:

* Bipolar or psychotic disorder
* Primary anxiety disorders without concomitant major depression as defined above
* Current significant suicidal ideation or behaviors require a higher level of care.
* Use of neuromodulation therapies (e.g., ECT, TMS, VNS) within the past 6 months.
* History of seizures, implanted cranial/ cardiac metal, or neurosurgery.
* Use of medications that significantly reduce seizure threshold
* Frequent/severe HA
* Personal history of head trauma, concussion, or TBI
* Catatonic or otherwise unable to perform the consent process
* Current alcohol or substance-use disorder (moderate-severe).
* Any non-uniformities in the skin under the electrode site, including eczema, severe rashes, hyperhidrosis, communicable skin disorders, sensitive skin (ex. eczema, severe rashes), blisters, open wounds, burns including sunburns, cuts or irritation (e.g. due to shaving), or other skin defects or lesions, as determined by clinical personnel
* Pregnancy (urine test required for women of childbearing potential).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Device-Related Serious Adverse Events | Up to 7 days
  Defined as events requiring hospitalization or emergency care during the stimulation period.
Number of Participants Completing All Scheduled Sessions Without Discontinuation | Completion of all planned stimulation sessions without dropout due to adverse effects.
  Up to 5 days
Mean Score on Adverse Event Questionnaire | Daily during treatment (Days 1-5)
  Average Likert-scale ratings of discomfort, headache, or skin irritation.

SECONDARY OUTCOMES:
Change in Depression Severity Score From Baseline to Post-Treatment | Baseline to Day 5
  Self-reported depression severity using a validated scale.
Change in Cognitive Function Score From Baseline to Post-Treatment | Baseline to Day 5
  Subjective cognitive performance measured via standardized instrument.
Change in Mindfulness Score From Baseline to Post-Treatment | Baseline to Day 5
  Self-reported mindfulness using a validated scale.
Change in Depression Severity Score From Baseline to 4-Week Follow-Up | Baseline to 4 weeks post-treatment
  Longitudinal assessment of symptom durability.
Electric Field Intensity in Target Brain Regions Based on MRI Modeling | Within 30 days of MRI scan
  Retrospective modeling of intracerebral current flow using structural MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Olash, MD, Study Director — Medical University of South Carolina
Locations (1):
- MUSC Brain Stimulation Lab, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (2):
  • Study Protocol (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/11/NCT07226011/Prot_000.pdf
  • Informed Consent Form (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/11/NCT07226011/ICF_001.pdf